CLINICAL TRIAL: NCT05371470
Title: Evaluation of Voice Analysis Technology in Detecting and Managing Depression and Anxiety in Patients Undergoing Cardiac Rehabilitation
Brief Title: Voice Analysis Technology to Detect and Manage Depression and Anxiety in Cardiac Rehabilitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-012982
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Infarction
Keywords: Cardiac Rehabilitation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cardiac rehabilitation plus voice analysis (Experimental): Subjects will complete 12 weeks of cardiac rehabilitation as per clinical care and utilize a voice analysis smartphone app.
  Interventions: Device: Ellipsis Health Voice Application
- Cardiac rehabilitation only (No Intervention): Subjects will complete 12 weeks of cardiac rehabilitation as per clinical care.

INTERVENTIONS:
Device: Ellipsis Health Voice Application — Smartphone application that utilizes voice biomarkers to assess for potential presence and severity of depression and anxiety
  Arms: Cardiac rehabilitation plus voice analysis

SUMMARY:
The purpose of this study is to learn if a voice analysis smartphone app which detects anxiety and depression could be used along with cardiac rehabilitation to improve results compared to cardiac rehabilitation alone.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. Enrolled in cardiac rehabilitation program to start within 3 months from hospital discharge
3. Owns a smartphone
4. Willing to download and use a smartphone app
5. Able to read, write, and speak English

Exclusion Criteria:

1. Cardiac transplant
2. Active substance use
3. Neurocognitive disorder
4. Active psychosis
5. Mania diagnosis
6. Active suicidality
7. Uncontrolled bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline, 12 weeks
  Measured using the self-reported Patient Health Questionnaire-9 (PHQ-9) to assess for major depressive disorder. Possible score range from 0 to 27, with higher scores indicating a worse outcome/greater severity of depressive symptoms.
Change in anxiety symptoms | Baseline, 12 weeks
  Measured using the self-reported Generalized Anxiety Disorder 7-Item Scale (GAD-7) that assesses anxiety symptoms. Possible score range from 0 to 21, with higher scores indicating a worse outcome/greater severity of anxiety symptoms.
Change in perceived stress | Baseline, 12 weeks
  Measured using the self-reported Perceived Stress Scale-14 (PSS-14), a 14 item questionnaire which assesses the degree to which situations in life are stressful within the last month. Each item is scored on a 5 point Likert scale from 0 (never) to 4 (very often), higher total scores indicate a worse outcome/greater severity of perceived stress.
Change in quality of life | Baseline, 12 weeks
  Measured using the self-reported abbreviated generic Quality of Life Scale developed through the World Health Organization (WHOQOL-BREF) questionnaire that assesses an individual's perceptions of their health and well-being within the last two weeks. Each item is scored on a 5 point Likert scale, higher scores indicate greater perceived quality of life.
Change in health behaviors | Baseline, 12 weeks
  Measured using the self-reported Current Health Behaviors (HB) questionnaire, a 13 item questionnaire which assesses behaviors and life circumstances during the last month. Each item is scored on a 10 point Likert scale, higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No